CLINICAL TRIAL: NCT04467931
Title: Association Between Angiotensin Converting Enzyme Inhibitor or Angiotensin Receptor Blocker Use and COVID-19 Severity and Mortality Among US Veterans
Brief Title: ACEI or ARB and COVID-19 Severity and Mortality in US Veterans
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency); University of Pennsylvania (Other); Wake Forest University Health Sciences (Other); University of Florida (Other); Johns Hopkins Bloomberg School of Public Health (Other); Boston University (Other); Northwestern University (Other); Edith Nourse Rogers Memorial Veterans Hospital (U.S. Federal Agency); Columbia University (Other); MedStar Georgetown University Hospital (Other)
Responsible Party: Principal Investigator, Adam Bress, Associate Professor, University of Utah
Other Study IDs: 00132408
Record Dates: First submitted 2020-07-06; First posted 2020-07-13 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; COVID
Keywords: angiotensin-converting enzyme inhibitor; angiotensin receptor antagonist; Veterans; antihypertensive medications
MeSH Terms: conditions — Hypertension | interventions — benazepril; Captopril; Enalapril; Fosinopril; Lisinopril; moexipril; Perindopril; Quinapril; Ramipril; trandolapril; azilsartan; candesartan; eprosartan; Irbesartan; Losartan; olmesartan; Telmisartan; Valsartan; Doxazosin; Prazosin; Terazosin; Acebutolol; Nebivolol; Atenolol; Betaxolol; Bisoprolol; Metoprolol; Pindolol; Penbutolol; Carvedilol; Labetalol; Nadolol; Propranolol; Timolol; Amlodipine; Felodipine; Isradipine; Nifedipine; Nicardipine; Nisoldipine; Diltiazem; Verapamil; Clonidine; Guanfacine; Guanabenz; Methyldopa; Reserpine; Hydralazine; Minoxidil; aliskiren; Spironolactone; Eplerenone; Bumetanide; Furosemide; Ethacrynic Acid; Torsemide; Amiloride; Triamterene; Bendroflumethiazide; Chlorothiazide; Chlorthalidone; Hydrochlorothiazide; Indapamide; Metolazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- 1.1 Outpatient SARS-CoV-2 Positive, ACEI/ARB vs non-ACEI/ARB: Among Veterans with treated hypertension and without compelling indications who test positive for SARS-CoV-2, compare all-cause hospitalization and all-cause mortality rates between current users of a range of doses of ACEI/ARB- vs. non-ACEI/ARB-based regimens.
  Interventions: Drug: ACEI/ARB; Drug: Non-ACEI/ARB
- 1.2 Outpatient SARS-CoV-2 Positive, ACEI vs. ARB: Among Veterans with treated hypertension who test positive for SARS-CoV-2, compare all-cause hospitalization and all-cause mortality rates between current users of a range of doses of ACEI- vs. ARB-based regimens.
  Interventions: Drug: ACEI; Drug: ARB
- 2.1 COVID-19 Hospitalized, ACEI/ARB vs non-ACEI/ARB: Among Veterans with treated hypertension and without compelling indications who are hospitalized for COVID-19, compare all-cause mortality rates between current users of a range of doses of ACEI/ARB- vs. non-ACEI/ARB-based regimens.
  Interventions: Drug: ACEI/ARB; Drug: Non-ACEI/ARB
- 2.2 COVID-19 Hospitalized, ACEI vs. ARB: Among Veterans with treated hypertension who are hospitalized for COVID-19, compare all-cause mortality rates between current users of a range of doses of ACEI- vs. ARB-based regimens.
  Interventions: Drug: ACEI; Drug: ARB

INTERVENTIONS:
Drug: ACEI/ARB — Veterans will be categorized as exposed to ACEI/ARB if they have one or more pharmacy fills for an oral ACEI or an ARB in the 90 days (± 14 days) prior to each Veteran's index date. Sacubitril/valsartan (Brand name: Entresto®) will be excluded from ARB exposures.
  Other Names: benazepril; captopril; enalapril; fosinopril; lisinopril; moexipril; perindopril; quinapril; ramipril; trandolapril; azilsartan; candesartan; eprosartan; irbesartan; losartan; olmesartan; telmisartan; valsartan
  Groups: 1.1 Outpatient SARS-CoV-2 Positive, ACEI/ARB vs non-ACEI/ARB; 2.1 COVID-19 Hospitalized, ACEI/ARB vs non-ACEI/ARB
Drug: Non-ACEI/ARB — Veterans will be categorized as exposed to a non-ACEI/ARB if they have one or more pharmacy fills for an oral non-ACEI or ARB medication in the 90 days (± 14 days) prior to each Veteran's index date and NO fills for an ACEI/ARB medication in the 90 days (± 14 days) prior to each Veteran's index date. Specific drug classes include: aldosterone receptor antagonist, beta-blocker, calcium channel blocker, centrally-acting drug, direct arterial vasodilator, direct renin inhibitor, thiazide diuretic, loop diuretic, and potassium sparing diuretic.
  Other Names: doxazosin; prazosin; terazosin; acebutolol; nebivolol; atenolol; betaxolol; bisoprolol; metoprolol; pindolol; penbutolol; carvedilol; labetalol; nadolol; propranolol; timolol; amlodipine; felodipine; isradipine; nifedipine; nicardipine; nisoldipine; diltiazem; verapamil; clonidine; guanfacine; guanabenz; methyldopa; reserpine; hydralazine; minoxidil; aliskiren; spironolactone; eplerenone; bumetanide; furosemide; ethacrynic acid; torsemide; amiloride; triamterene; bendroflumethiazide; chlorothiazide; chlorthalidone; hydrochlorothiazide; indapamide; metolazone
  Groups: 1.1 Outpatient SARS-CoV-2 Positive, ACEI/ARB vs non-ACEI/ARB; 2.1 COVID-19 Hospitalized, ACEI/ARB vs non-ACEI/ARB
Drug: ACEI — Veterans will be categorized as exposed to an ACEI if they have one or more pharmacy fills for an oral ACEI in the 90 days (± 14 days) prior to each Veteran's index date and NO fills for an oral ARB in the 90 days (± 14 days) prior to each Veteran's index date.
  Other Names: benazepril; captopril; enalapril; fosinopril; lisinopril; moexipril; perindopril; quinapril; ramipril; trandolapril
  Groups: 1.2 Outpatient SARS-CoV-2 Positive, ACEI vs. ARB; 2.2 COVID-19 Hospitalized, ACEI vs. ARB
Drug: ARB — Veterans will be categorized as exposed to an ARB if they have one or more pharmacy fills for an oral ACEI in the 90 days (± 14 days) prior to each Veteran's index date and NO fills for an oral ACEI in the 90 days (± 14 days) prior to each Veteran's index date. Sacubitril/valsartan (Brand name: Entresto®) will be excluded from ARB exposures.
  Other Names: azilsartan; candesartan; eprosartan; irbesartan; losartan; olmesartan; telmisartan; valsartan
  Groups: 1.2 Outpatient SARS-CoV-2 Positive, ACEI vs. ARB; 2.2 COVID-19 Hospitalized, ACEI vs. ARB

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus responsible for COVID-19, enters type II pneumocytes using angiotensin-converting enzyme 2 (ACE2). It is unclear whether ACE inhibitors (ACEIs) and angiotensin receptor blockers (ARBs) increase, decrease, or have no significant effect on ACE2 expression or activity. Therefore, ACEI and ARB may be harmful, beneficial, or have no impact on Coronavirus Disease 2019 severity and mortality. The Specific Aims of this observational study are: (1) Among SARS-CoV-2-positive outpatients, compare all-cause hospitalization and mortality rates between: 1.1 Current users of a range of doses of ACEI/ARB- vs. non- ACEI/ARB-based regimens, and 1.2 Current users of a range of doses of ACEI- vs. ARB-based regimens, and (2) Among those hospitalized for COVID-19, compare all-cause mortality between: 2.1 Current users of a range of doses of ACEI/ARB- vs. non- ACEI/ARB-based regimens, and 2.2 Current users of a range of doses of ACEI- vs. ARB-based regimens.

DETAILED DESCRIPTION:
The Coronavirus Disease 2019 (COVID-19) pandemic has killed >129,000 Americans as of June 30, 2020. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus responsible for COVID-19, enters type II pneumocytes using angiotensin-converting enzyme 2 (ACE2). ACE inhibitors (ACEIs) and angiotensin receptor blockers (ARBs) may increase ACE2 expression. Theoretically, if ACEI/ARB use increases ACE2 expression in the lungs, ACEI/ARBs could promote SARS-CoV-2 entry into type II pneumocytes and worsen COVID-19 infection. In contrast, other evidence suggests that ACEI/ARBs may mitigate virus-induced inflammatory responses in the lungs by upregulating ACE2-mediated generation of the vasodilator and anti-inflammatory protein angiotensin-(1-7), thereby preventing tissue damage. Few data exist on the direction or magnitude of the association between ACEI/ARB use and COVID-19 severity, and whether these associations differ between ACEIs and ARBs. Because ACEI/ARBs are among the most commonly used prescription medications, it is critical to determine if ACEI/ARB users have a differential risk of more severe COVID-19 infection compared to non-users. The objective of this study is to reduce morbidity and mortality of the COVID-19 pandemic by generating timely evidence on the direction and magnitude of the association between ACEI/ARB use and COVID-19 severity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test in the outpatient setting (Aim 1) or hospitalized for COVID-19 (Aim 2)
* Meet continuous enrollment criteria (≥1 inpatient or any outpatient encounter in each of the two, six-month periods during the 365 days prior to the index date)
* Do not have data inconsistencies (test patients, not Veterans, multiple death dates in data, or not alive on index date)
* Diagnosed with hypertension at any point prior to the index date
* Had at least one prescription dispensed for an antihypertensive medication in the 90 days prior to the index date

Exclusion Criteria:

* Aim 1.1 and 2.1 (ACEI/ARB vs. non-ACEI/ARB comparison): diagnosed with a compelling indication for ACEI/ARB at any point prior to the index date (i.e., diabetes, stroke, chronic kidney disease, heart failure with reduced ejection fraction, or coronary heart disease)
* Aim 1.2 and 2.2 (ACE vs. ARB comparison): prescription fills for both an ACEI and an ARB in the 90 days prior to the index date; no prescription fill for an ACEI or an ARB in the 90 days prior to the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim 1: Positive test for SARS-CoV-2 in the outpatient setting, diagnosed with hypertension prior to the index date, and be treated with an antihypertensive in the 90 days prior to the index date.
  Aim 2: Hospitalized for COVID-19, diagnosed with hypertension prior to the index date, and be treated with an antihypertensive in the 90 days prior to the index date.
  ACEI/ARB vs. non-ACEI/ARB analyses (aims 1.1 and 2.1): Do not have compelling indications that would warrant preferential treatment with an ACEI or an ARB (i.e., diabetes, stroke, chronic kidney disease, heart failure with reduced ejection fraction, or coronary heart disease).
  ACEI vs. ARB analyses (aims 1.2 and 2.2): Not concomitantly treated with an ACEI and an ARB in the 90 days prior to the index date, and must be treated with at least an ACEI or an ARB in the 90 days prior to the index date.
Sampling Method: Non-Probability Sample
Enrollment: 22213 (Actual)
Dates: Start 2020-01-19 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
All-Cause-Hospitalization or All-Cause Mortality | Through study completion (October 21, 2020).
  For outpatient Veterans with a positive SARS-CoV-2 test (Aims 1.1 and 1.2), the primary outcome is a composite of time to all-cause hospitalization or all-cause mortality.
All-Cause Mortality | Through study completion (October 21, 2020).
  For Veterans hospitalized with COVID-19 (Aims 2.1 and 2.2), the primary outcome is time to all-cause mortality.

SECONDARY OUTCOMES:
ICU admission | Through study completion (October 21, 2020).
  For aims 1 and 2, a secondary outcome will be time to intensive care unit (ICU) admission.
Mechanical ventilation | Through study completion (October 21, 2020).
  For aim 2, a secondary outcome will be time to mechanical ventilation.
Dialysis | Through study completion (October 21, 2020).
  For aim 2, a secondary outcome will be time to in-hospital dialysis.

OTHER OUTCOMES:
Negative control outcomes (Gastrointestinal bleed or urinary tract infection) | Through study completion (October 21, 2020).
  Time to first occurrence of gastrointestinal bleed or urinary tract infection. This will be a negative control outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Bress, PharmD, MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Derington CG, Cohen JB, Mohanty AF, Greene TH, Cook J, Ying J, Wei G, Herrick JS, Stevens VW, Jones BE, Wang L, Zheutlin AR, South AM, Hanff TC, Smith SM, Cooper-DeHoff RM, King JB, Alexander GC, Berlowitz DR, Ahmad FS, Penrod MJ, Hess R, Conroy MB, Fang JC, Rubin MA, Beddhu S, Cheung AK, Xian W, Weintraub WS, Bress AP. Angiotensin II receptor blocker or angiotensin-converting enzyme inhibitor use and COVID-19-related outcomes among US Veterans. PLoS One. 2021 Apr 23;16(4):e0248080. doi: 10.1371/journal.pone.0248080. eCollection 2021. PMID 33891615

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04467931/Prot_SAP_000.pdf